CLINICAL TRIAL: NCT06489262
Title: Efficacy Trial of Healthy Together "Juntos": A Family-based Digital Lifestyle Intervention for Hispanic Adolescents and Their Parents
Brief Title: Efficacy Trial of Healthy Together ("Juntos")
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sara StGeorge, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20231382; R01CA289519 (NIH)
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Activity, Motor; Diet, Healthy
Keywords: Hispanic, family, digital health, obesity prevention, physical activity, nutrition
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Together ("Juntos") (Experimental): Participants will receive the Healthy Together ("Juntos") digital intervention. The six-month intervention includes an "intensive" phase comprised of eight modules and coaching sessions delivered in the first three months and a "maintenance phase" comprised of three modules and coaching sessions delivered in the subsequent three months.
  Interventions: Behavioral: Healthy Together ("Juntos")
- Control (No Intervention): This group will receive a digital standard of care - a list of publicly available lifestyle apps and websites that they may access at their discretion.

INTERVENTIONS:
Behavioral: Healthy Together ("Juntos") — Parent-adolescent dyads will log in to a secured website for six months. The intervention will be delivered primarily through smartphones and will include didactic content on healthy lifestyle behaviors (for parents/adolescents), family behavior change content for setting weekly goals and self-monitoring health behaviors (for parents/adolescents), and positive parenting content (for parents only), all of which were developed in accordance with participant feedback based on formative intervention development work. In addition, and to increase participant compliance/reduce attrition often observed in digital health interventions, human support ("supportive accountability") will be provided. Specifically, each family will be assigned a "coach" who will use video conferencing software to engage in approximately weekly (during the first 3 months), and monthly (during the following 3 months) 20-30-minute sessions regarding the family's progress throughout the intervention period.
  Arms: Healthy Together ("Juntos")

SUMMARY:
The purpose of this study is to assess the efficacy of a family-based digital (web and mobile phone-based) program known as Healthy Together ("Juntos") in preventing increases in body mass index and improving moderate-to-vigorous physical activity, diet quality, and percentage body fat among Hispanic adolescents.

ELIGIBILITY:
Inclusion Criteria:

Adolescent

1. Lives with participating biological parent or legal guardian;
2. Self-identifies as Hispanic;
3. Is between the ages of 12-15years old;
4. Has access to a smartphone;
5. Does not meet recommendations for physical activity as determined by a validated 2-item screener;
6. Does not meet recommendations for daily fruit and vegetable intake (proxy for diet quality) as determined by a validated 2-item screener;
7. Exceeds recommendations for screen time (proxy for sedentary behavior) as determined by a validated 6-item screener

Parent

1. Is the biological parent or legal guardian of and lives with the adolescent;
2. Self-identifies as Hispanic;
3. Has access to a smartphone;

Exclusion Criteria:

Adolescent

1. Has BMI <5th (underweight) or ≥95th percentile (obesity);
2. Has a parent-reported chronic medical condition (e.g., type 2 diabetes) that requires more intensive intervention;
3. Has parent-reported responses on a physical activity readiness questionnaire (PAR-Q) that indicates a serious health issue, and a physician does not approve participation;
4. Has a parent-reported cognitive or developmental delay (e.g., Down Syndrome) that may interfere with understanding program materials.

Parent

1. Provides PAR-Q responses that indicate a serious health issue and a physician does not approve participation;
2. Reports family plans to move out of South Florida during the study follow-up period

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) in adolescents | Baseline and up to 12 months
  Will be measured in kg/m^2

SECONDARY OUTCOMES:
Change in Moderate-to-Vigorous Physical Activity (MVPA) in adolescents | Baseline and up to 12 months
  Will be measured using an Actigraph (counts/seconds (Moderate=757-1111 counts/15-seconds and vigorous>1200 counts/15-seconds))
Change in Diet Quality in adolescents measured by National Cancer Institute (NCI) Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool | Baseline and up to 12 months
  Healthy Eating Index scores range from 0-100, higher scores indicate a higher quality diet
Change in Percentage of Body Fat in adolescents | Baseline and up to 12 months
  Measured in percentage
Change in Body Mass Index (BMI) in parents | Baseline and up to 12 months
  Will be measured in kg/m^2
Change in Moderate-to-Vigorous Physical Activity (MVPA) in parents | Baseline and up to 12 months
  Will be measured using an Actigraph (in counts/minutes (Moderate=2690-6166 - counts/minute; vigorous≥6167 counts/min))
Change in Diet Quality in parents measured by National Cancer Institute (NCI) Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool | Baseline and up to 12 months
  Healthy Eating Index scores range from 0-100, higher scores indicate a higher quality diet
Change in Percentage of Body Fat in parents | Baseline and up to 12 months
  Measured in percentage
Change in Parenting Practices measured by the Parental involvement Scale | Baseline and up to 12 months
  Measured by parental involvement subscale of the Parenting Practices measure (4-point Likert scale, higher scores indicate higher parental involvement; parent and adolescent report)
Change in Communication measured by Parent Adolescent Communication Scale | Baseline and up to 12 months
  Measured by the Parent-Adolescent Communication Scale (5-point Likert scale, higher scores indicate more positive communication; parent and adolescent report)
Change in Health-related Positive Parenting Practices measured by the Parenting Strategies for Eating and Activity Scale | Baseline and up to 12 months
  Measured by the Parenting Strategies for Eating and Activity Scale (5-point Likert scale, higher scores indicate more use of parent strategies for heathy eating and activity; parent and adolescent report)

CONTACTS AND LOCATIONS:
Overall Officials: Sara St George, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No